CLINICAL TRIAL: NCT03902509
Title: A Randomized, Controlled, Multi-site Study About Safety and Efficacy of Pirfenidone to Treat Grade 2 or Grade3 Radiation-induced Lung Injury.
Brief Title: A Study About Safety and Efficacy of Pirfenidone to Treat Grade 2 or Grade3 Radiation-induced Lung Injury.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-F647-201901
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2023-12

CONDITIONS: Radiation-induced Lung Injury
Keywords: pirfenidone
MeSH Terms: interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pirfenidone (Experimental): pirfenidone + basic treatment
  Interventions: Drug: Pirfenidone; Drug: basic treatment
- Controll (Other): with basic treatment and without pirfenidone treatment
  Interventions: Drug: basic treatment

INTERVENTIONS:
Drug: Pirfenidone — pirfenidone capsule made in China
  Arms: Pirfenidone
Drug: basic treatment — glucocorticoid and expectant treatment etc.

SUMMARY:
Using Pirfenidone to treat Grade 2 or Grade3 radiation-induced lung injury, and observe the efficacy and safety of the drug.

DETAILED DESCRIPTION:
The study is a randomized, controlled, multi-site clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old (including 18 and 75 years);
2. clinically diagnosed grade 2 or 3 radiation-induced lung injury;
3. the course of radiation-induced lung injury is less than 2 months;
4. ECOG 0-2;
5. the expected survival time is more than 6 months;
6. the functional level of major organs meets the following standards: ANC≥3.0×109/L，PLT≥100×109/L，Hb≥90g/L, TBIL、BUN and Cr≤1.5×ULN， ALT、AST≤2.0×ULN
7. capable of eating solid food upon enrollment;
8. subjects will voluntarily participate in this study and sign the informed consent.

Exclusion Criteria:

1. have a history of chronic bronchial acute attack or severe pulmonary heart disease;
2. pneumonectomy;
3. tumor progression;
4. severe pulmonary infection;
5. creatinine clearance rate < 30ml/min, severe renal disease or need dialysis;
6. concomitant with other serious diseases: for example, myocardial infarction within 6 months, uncontrolled diabetes, etc., were considered not suitable for the participants in the study;
7. patients with active peptic ulcer;
8. pregnant women and patients with mental illness;
9. participating in clinical trials of other drugs within 3 months;
10. the investigator determined that subject was not suitable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
DLco% change | Week 4, 8,16, and 24
  Compare DLco% from basement to the end of treatment

SECONDARY OUTCOMES:
The grade change of radiation-induced lung injury | Week 4, 8,16, and 24
The score change of CT | Week 4, 8,16, and 24
Increase of effective lung volume | Week 4, 8,16, and 24
The grade change of Cough, Dyspnea and Fever | Week 4, 8,16, and 24

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hou Z, Dong B, Yao Q, Chen H, Shao Q, Li M, Wang J, Chen K, Zhu Z, Peng F, Wei S, Hu X, Li J, Liu M, Xu B, Zheng S, Bi N, Zheng S, Xu Q, Chen B, Wu C, Li R, Chen W, Liu X, Tian Y, Li X, Guo S, Zhao L, Zhu Y, Cai L, Li Q, Li L, Zhang H, Hu C, Wang L, Li Q, Chen B, Chen M. Pirfenidone for grade 2 and grade 3 radiation-induced lung injury: a multicentre, open-label, randomised, phase 2 trial. Lancet Oncol. 2025 Dec;26(12):1552-1562. doi: 10.1016/S1470-2045(25)00515-7. Epub 2025 Nov 6. PMID 41207313